CLINICAL TRIAL: NCT04918563
Title: Investigation of the Endothel Dependent and Independent Vasodilatation in Human Gingiva: Comparison of the Effect of NO and ACH
Brief Title: Endothelium Dependent and Non-dependent Vasodilatation in Human Gingiva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Vag Janos, associate professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1/2020
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Vasodilatation; Oral Soft Tissue Conditions
Keywords: spreading vasodilatation; gingial microcirculation; LSCI
MeSH Terms: conditions — Aneurysm | interventions — Nitroglycerin; Acetylcholine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nitroglycerin (Active Comparator): NO donor (Nitropohl) vs pgysiological saline
  1mg/ml nitorhlycerin
  Interventions: Drug: Nitroglycerin
- acethylcholine (Active Comparator): 10 mg/ml acetylcholine vs physiological saline
  Interventions: Drug: Acetylcholine

INTERVENTIONS:
Drug: Nitroglycerin — Vasodilatator solution is dropped on the labial surface on the lateral incisor, so it can penetrate through the sulcus.
  Arms: nitroglycerin
Drug: Acetylcholine — Vasodilatator solution is dropped on the labial surface on the lateral incisor, so it can penetrate through the sulcus.
  Other Names: Ach
  Arms: acethylcholine

SUMMARY:
The aim of this study is to compare the endothelim-dependent and non-dependent vasodilatation between genders in the human gingiva.

DETAILED DESCRIPTION:
Gender differences were observed in studies according to gingival microcirculation between physiological circumstances and during wound healing as well.

For blood flow measurement Laser Spackle Contrast Imaging is a reliable tool. It has good reproducibility, it doesn't get in touch with the measured surface, it's easy to use and it can measure on a bigger surface in same time.

Two wells were fabricated on the labial surface of the right lateral incisor (test tooth) and on the labial surface of the left central incisor (control tooth). These wells are opened towards the high-prermeability gingival sulcus, so the dropped solutions nitroglycerine vs physiological saline or nitroglycerine vs physiological saline can esasily penetrate to the gingival tissues. After applying the solutions, the blood flow was monitored fot 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* general health
* minimum 5 mm keratinized gingiva at the upper front teeth
* good oral hygiene

Exclusion Criteria:

* pregnancy and breast-feeding
* smoking
* medication
* insufficient marginal integrity
* periodontitis
* caries

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Blood flow change after applying the test solutions | 20 minutes
  The change in blood flow will be measeured after applying the test solutions.

SECONDARY OUTCOMES:
Comparison the change in blood flow between the two solutions | 30 minutes
  The blood flow values will be evaluated after each applied solutions.
Comparison the change in blood flow in genders | 20 minutes
  The maximal blood flow changes assessed in primary outcome will be split into two groups based on gender. The change will be compared between males and females.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Department of Conservative Dentistry, Budapest, Hungary

REFERENCES:
- [Derived] Vag J, Nagy TL, Mikecs B. Sex-related differences in endothelium-dependent vasodilation of human gingiva. BMC Oral Health. 2022 May 13;22(1):177. doi: 10.1186/s12903-022-02186-2. PMID 35562729